CLINICAL TRIAL: NCT03531801
Title: Pressure-induced Referred Pain is More Expansive in Individuals With a Recovered Non-painful Fracture
Brief Title: Referred Pain Areas in Subjects With a Recovered Radius Fracture
Status: Completed | Type: Observational
Sponsor: Universidad San Jorge (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Víctor Doménech, Lecturer and Researcher at Universidad San Jorge, Universidad San Jorge
Other Study IDs: PI16/094
Record Dates: First submitted 2018-04-25; First posted 2018-05-22 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Radius Fractures
Keywords: Referred pain; pressure algometry; pain mapping
MeSH Terms: conditions — Radius Fractures; Pain, Referred

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recovered fracture group: The interventions will be conducted on both groups, on two experimental (approximately 45 minutes per session) sessions separated by 24 hours.Pressure algometry consists of measuring pressure pain thresholds at three bilateral muscle sites.Mapping referred pain areas consists of recording on an electronic body chart the area of pain induced by 60s pressure stimulation at 1.2 times the force needed to reach the pressure pain threshold, exerted on the extensor carpi radialis and the infraspinatus muscles.As group-differences can be attenuated at baseline but emerge on a sensitized (exercise-induced soreness) state, these procedures are performed at baseline and 24 hours after evoking exercise-induced muscle soreness. For further clarification see our recent publication PMID:29608510
  Interventions: Other: Pressure algometry and mapping referred pain areas
- Control group: This group will receive the same intervention than the recovered fracture group
  Interventions: Other: Pressure algometry and mapping referred pain areas

INTERVENTIONS:
Other: Pressure algometry and mapping referred pain areas — The described procedures are tested at baseline and 24 hours after exercise-induced muscle soreness conditions.
  Other Names: Delayed onset muscular soreness

SUMMARY:
The purpose of the present study is to investigate pressure algometry and pressure-induced referred pain areas in pain free individuals with a history of distal radius fracture (fully recovered) compared with age and gender matched healthy controls without history of fracture. It is hypothesized that individuals with a recovered radius fracture will have a facilitated referred pain patter towards the wrist but normal pressure pain sensitivity.

DETAILED DESCRIPTION:
Musculoskeletal injuries, nociception and pain can increase the sensitivity of the central pain mechanisms, which can be extended even after tissue recovery. However, little is known about the status of these central pain mechanisms once subjects are fully recovered from the tissue injury and pain. This information would help to explain pain conditions in which recurrence of the pain episodes is common (e.g low back pain or shoulder pain).

Pressure-pain thresholds have been widely used in pain research to test the sensitivity of the pain system. Additionally, referred pain has been shown as a valid biomarker for the sensitization of the pain system.

The aim of the present study is to investigate pressure pain sensitivity and referred pain patterns of individuals with a history of recovered fracture, compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of distal radius fracture without pain at the moment of the study.

Exclusion Criteria:

* Subjects with symptoms (e.g pain), functional limitations, history of other fractures in the upper limb or any other pathology.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with a history of distal radius fracture without pain at the moment of the study or any physical sequelae derived from the fracture.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
A change in the area of referred rain | 24 hours (two experimental sessions separated by 24h).
  This outcome measure corresponds to the difference or change in the size and distribution of the pressure-induced referred pain area, between the two experimental sessions.

SECONDARY OUTCOMES:
A change in pressure-pain thresholds | 24 hours (two experimental sessions separated by 24h).
  This secondary outcome measure corresponds to the force required to produce a MINIMAL pain(1 out of 10 on a 0-10 visual analogue scale)

CONTACTS AND LOCATIONS:
Overall Officials: Víctor Doménech-García, MSc, Principal Investigator — Universidad San Jorge
Locations (1):
- Universidad San Jorge, Villanueva de Gállego, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan at the moment